CLINICAL TRIAL: NCT01660542
Title: An Open-label, Multi-center Phase Ⅳ Trial to Evaluate the Efficacy and Safety of Sequential Neoadjuvant Chemotherapy With Docetaxel(Monotaxel®) After Doxorubicin Plus Cyclophosphamide Combination Chemotherapy in Locally Advanced Breast Cancer
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4-2011-0068
Record Dates: First submitted 2012-08-05; First posted 2012-08-08 (Estimated); Last update posted 2016-11-01 (Estimated); Status verified 2016-10

CONDITIONS: Locally Advanced Breast Cancer
MeSH Terms: interventions — Neoadjuvant Therapy; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- doxorubicin/cyclophosphamide (Experimental): Neoadjuvant Chemotherapy with Docetaxel(Monotaxel®) after Doxorubicin plus Cyclophosphamide
  Interventions: Drug: Neoadjuvant Chemotherapy with Docetaxel

INTERVENTIONS:
Drug: Neoadjuvant Chemotherapy with Docetaxel — Doxorubicin 60 mg/m2 plus cyclophosphamide 600 mg/m2 (day 1), IV (in the vein), every 21 days, a total of 4 cycles -> Docetaxel 100 mg/m2 (day 1) IV, every 21 days, a total of 4 cycles

SUMMARY:
This is a multicenter, open-label, phase IV trial to assess the efficacy and safety of sequential neoadjuvant chemotherapy with 4 cycles of doxorubicin/cyclophosphamide followed by 4 cycles of docetaxel(Monotaxel®) in patients with breast cancer of ≥5cm in size or cytologically confirmed axillary lymph nodes metastasis.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically proven invasive breast cancer - the primary tumor size is at least 5cm or cytologically proven axillary node metastasis
2. no evidence of systemic metastasis pathologically or radiologically
3. age at the time of diagnosis between 20 and 70 years
4. patients with previously untreated primary breast cancer including chemotherapy
5. general performance status with ECOG 0-2
6. sufficient hematopoietic function (absolute neutrophil count of ≥ 1,500/mm3, platelet count of ≥ 100,000/mm3, and hemoglobin of ≥ 10 g/dL)
7. sufficient renal function (serum creatinine level of ≤ 1.5 mg/dL)
8. sufficient liver function (total serum bilirubin level ≤ 1.5 times the upper normal limit; serum AST and ALT levels ≤ 1.5 times the upper normal limit; and serum alkaline phosphatase level ≤ 1.5 times the upper normal limit)
9. sufficient cardiac function (normal electrocardiography within 1 month or LVEF>50% by echocardiography or MUGA scan within 3 months)
10. patients who agree to enroll this clinical trial and sign the written informed consent voluntarily

Exclusion Criteria:

1. patients with evidence of distant metastases
2. patients with other previous malignancy except breast cancer
3. pregnant (positive hCG test 1 week before registration) or lactating patient
4. uncontrolled serious infection
5. patients with psychiatric disease or epilepsy
6. patients with clinically severe cardiac disease within 6 months such as atrial or ventricular arrhythmia, congestive heart failure, myocardial infarction, or unstable angina
7. male breast cancer
8. patients with poor general condition who are not able to understand or sign the written informed consent

Ages: 20 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2011-04; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Pathologic Complete Response | 26 weeks after the first administration of neoadjuvant chemotherapy with doxorubicin/cyclophosphamide regimens
  Pathologic complete response is defined as the disappearance of all invasive cancer in the postsurgical breast and lymph node specimens after completion of neoadjuvant chemotherapy. Only residual intraductal carcinoma in the postsurgical breast specimen after neoadjuvant chemotherapy is also considered as the achievement of pathologic complete response.

CONTACTS AND LOCATIONS:
Locations (1):
- Severance hospital, Seoul, Seoul, South Korea